CLINICAL TRIAL: NCT06171074
Title: A Multicenter, Single Arm Phase II Clinical Study Evaluating the Efficacy of CM310 Recombinant Humanized Monoclonal Antibody Injection in Patients With Seasonal Allergic Rhinitis
Brief Title: Study of CM310 in Subjects With Seasonal Allergic Rhinitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310-107105
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental): CM310, Subcutaneous injection
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310 injection

SUMMARY:
This study is a multicenter, single arm phase II clinical study mainly evaluating the efficacy of CM310 in patients with seasonal allergic rhinitis.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a non infectious chronic inflammatory disease of the nasal mucosa that is mainly mediated by immunoglobulin E (IgE) in atopic individuals exposed to allergens.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65.
* Understand the study and sign the Informed Consent Form voluntarily.
* Take effective contraception measures throughout the study period.

Exclusion Criteria:

* Used other investigational drugs.
* Allergies to drugs with IL-4Rα monoclonal antibody or drug components of CM310.
* Plan to participate in other studies during this clinical trial.
* With malignant or benign tumors of the nasal cavity.
* Other reasons the researcher believes that the subject is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline mean of daily retrospective total nasal of symptom score (rTNSS) | Up to week 12
  The total score of nasal symptoms (TNSS) is the sum of four symptom scores: runny nose, nasal congestion, nasal itching, and sneezing, with each symptom scoring from 0 to 3 points.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tong-Ren hospital, Beijing, China